CLINICAL TRIAL: NCT05433922
Title: A Multicenter, Single-arm Clinical Study of the Efficacy and Safety of CSA in Combination With Avatrombopag for the Treatment of Primary Treatment of Severe Aplastic Anemia in the Elderly
Brief Title: Efficacy and Safety of CSA and Avatrombopag for the Treatment of SAA in the Elderly
Acronym: SAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Fengkui Zhang, Director of Anemia Treatment Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fkzhang
Record Dates: First submitted 2022-06-11; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Severe Aplastic Anemia
Keywords: Avatrombopag; Aplastic Anemia; elderly; sever
MeSH Terms: conditions — Anemia, Aplastic | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CSA + Avatrombopag (Experimental): cyclosporine 3 mg/kg orally in two doses, with cyclosporine trough concentrations maintained at 200-250 ng/ml for 3 months to achieve maximum efficacy and then tapered by 25 mg every 3 months; Avatrombopag: two dosing groups, 40 mg orally once daily and 60 mg orally once daily, for a total of 24 weeks.If the 40 mg dose group trial meets the desired trial objectives, the 60 mg dose group trial will not be conducted.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — cyclosporine in combination with Avatrombopag to treat
  Other Names: CSA

SUMMARY:
This is a multicenter, single-arm clinical study. The objective was to evaluate the efficacy and safety of CSA in combination with Avatrombopag in elderly patients with very/sever aplastic anemia treated for the first time. The design was: cyclosporine 3 mg/kg orally in two divided doses, with cyclosporine trough concentrations maintained at 200-250 ng/ml for 3 months to achieve maximum efficacy, and Avatrombopag, which was administered in two dose groups, 40 mg orally once daily and 60 mg orally once daily, for a total of 24 weeks. Forty patients are expected to be enrolled in each dose group, and a total of 80 patients are expected to be enrolled if both dose groups are conducted. Evaluation endpoint: OR rate at 24 weeks of treatment.

DETAILED DESCRIPTION:
This is a multicenter, single-arm clinical study to evaluate the efficacy and safety of CSA combined with Avatrombopag. The patients are older than 60 years with diagnosis of very sever/sever aplastic anemia(V/SAA) without treatment before.

CSA is started at 3 mg/kg orally in two doses. Concentrations maintained at 200-250 ng/ml to achieve maximum efficacy and then tapered by 25 mg every 3 months; Avatrombopag: two dosing groups, 40 mg orally once daily and 60 mg orally once daily, for a total of 24 weeks；Each dose group is expected to include 40 patients each. If the 40 mg dose group trial meets the desired trial objectives, the 60 mg dose group trial will not be conducted, and if the 40 mg dose group does not meet the desired trial objectives, the 60 mg dose group trial will be continued. A total of 80 patients were expected to be included if both dose groups were conducted.Overall response rate at 24 weeks of treatment and adverse events are the evaluation endpoint.Secondary study endpoints were: CRR and ORR at 12 and 52 weeks of treatment, CRR at 24 weeks, survival, and clonal evolution in follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. elderly patients with V/SAA with a definite diagnosis.
2. age greater than 60 years, male or female.
3. Subjects must complete all screening assessments as outlined in the trial protocol.
4. Able to swallow or administer the drug orally.
5. Cannot tolerate or refuse ATG therapy.
6. No prior treatment with cyclosporine, tacrolimus or hormones or treatment for no more than 2 weeks.
7. No prior application of TPO receptor agonists (including Thrombopoietin, Eltrombopag, Hetrombopag, etc.) or application of TPO receptor agonists for treatment with ≤ 5 total doses and ≤ 7 days of TPO receptor agonist drugs such as Eltrombopag, Hetrombopag, etc.
8. Informed consent must be signed prior to the start of all specific study procedures, in consideration of the patient's condition, or by a member of the patient's immediate family if the patient's signature is not conducive to the treatment of the condition.

Exclusion Criteria:

No subject shall be enrolled in this study if he/she meets any of the following criteria.

1. known diagnosis of congenital hematopoietic failure disorders (e.g. Fanconi anemia) and other causes of allogeneic cytopenias and bone marrow hypoproliferative disorders (e.g. hemolytic PNH, hypoproliferative MDS/AML, autoantibody-mediated allogeneic cytopenias, etc.);
2. Patients with uncontrolled bleeding and/or infection despite standard treatment.
3. patients with previous history of hematopoietic stem cell transplantation;
4. previous history of thrombosis.
5. Patients with concurrent malignancy or potential cancer on immunosuppressive therapy.
6. Those who are considered unsuitable for enrollment by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
OR rate at 24 weeks of treatment | 24 weeks of treatment
  Percentage of the total number of patients receiving treatment who received a response at 24 weeks of treatment
Incidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading at 24 weeks of treatment | 24 weeks of treatment
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation at 24 weeks | 24 weeks of treatment
  % of patients with transformation to PNH or MDS,AML, or other disease

SECONDARY OUTCOMES:
OR rate and CR rate at 12 weeks | 12 weeks of treatment
  Percentage of patients who received a response and who receive a complete response at 12 weeks of treatment
Incidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading at 12 weeks | 12 weeks of treatment
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation at 12 weeks | 12 weeks of treatment
  % of patients with transformation to PNH or MDS,AML, or other disease at 12 weeks

OTHER OUTCOMES:
OR rate and CR rate at 52 weeks | 52 weeks of treatment
  Percentage of patients who received a response and who receive a complete response at 52 weeks of treatment
Incidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading at 52 weeks | 52 weeks of treatment
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation at 52 weeks | 52 weeks of treatment
  % of patients with transformation to PNH or MDS,AML, or other disease at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, doctor, Study Director — Anemia Treatment Center; Lei Ye, doctor, Principal Investigator — Anemia Treatment Center
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
You can ask for the researcher after completing the experiment
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Follow-up and publication of the paper are planned for December 2024
Access Criteria: After the paper is written and published

REFERENCES:
- [Result] Young NS, Kaufman DW. The epidemiology of acquired aplastic anemia. Haematologica. 2008 Apr;93(4):489-92. doi: 10.3324/haematol.12855. No abstract available. PMID 18379007
- [Result] Red Blood Cell Disease (Anemia) Group, Chinese Society of Hematology, Chinese Medical Association. [Chinese expert consensus on the diagnosis and treatment of aplastic anemia (2017)]. Zhonghua Xue Ye Xue Za Zhi. 2017 Jan 14;38(1):1-5. doi: 10.3760/cma.j.issn.0253-2727.2017.01.001. No abstract available. Chinese. PMID 28219216
- [Result] Contejean A, Resche-Rigon M, Tamburini J, Alcantara M, Jardin F, Lengline E, Ades L, Bouscary D, Marcais A, Lebon D, Chabrot C, Terriou L, Barraco F, Banos A, Bussot L, Cahn JY, Hirsch P, Maillard N, Simon L, Fornecker LM, Socie G, de Latour RP, de Fontbrune FS. Aplastic anemia in the elderly: a nationwide survey on behalf of the French Reference Center for Aplastic Anemia. Haematologica. 2019 Feb;104(2):256-262. doi: 10.3324/haematol.2018.198440. Epub 2018 Sep 27. PMID 30262561
- [Result] Scheinberg P. Activity of eltrombopag in severe aplastic anemia. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):450-456. doi: 10.1182/asheducation-2018.1.450. PMID 30504345
- [Result] Townsley DM, Scheinberg P, Winkler T, Desmond R, Dumitriu B, Rios O, Weinstein B, Valdez J, Lotter J, Feng X, Desierto M, Leuva H, Bevans M, Wu C, Larochelle A, Calvo KR, Dunbar CE, Young NS. Eltrombopag Added to Standard Immunosuppression for Aplastic Anemia. N Engl J Med. 2017 Apr 20;376(16):1540-1550. doi: 10.1056/NEJMoa1613878. PMID 28423296